CLINICAL TRIAL: NCT00834678
Title: Phase I/II Study of Bendamustine and Erlotinib for Metastatic or Locally Advanced Triple Negative Breast Cancer
Brief Title: Bendamustine and Erlotinib in Treating Patients With Stage IIIB, Stage IIIC, or Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08164; NCI-2011-03164 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2009-01-31; First posted 2009-02-03 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; estrogen receptor-negative breast cancer; HER2-negative breast cancer; progesterone receptor-negative breast cancer; triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Triple Negative Breast Neoplasms | interventions — Bendamustine Hydrochloride; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bendamustine and Erlotinib (Experimental): Bendamustine 100 or 120 mg/m2 IV on days 1 and 2 and erlotinib 100 or 150 mg po on days 5 - 21 of each 28 day cycle.
  Interventions: Drug: bendamustine; Drug: erlotinib; Drug: Maintenance erlotinib

INTERVENTIONS:
Drug: bendamustine — 100 or 120 mg/m2 IV on days 1 and 2
  Other Names: Ribomustin; Treanda; SDX- 105
Drug: erlotinib — 100 or 150 mg po on days 5 - 21 of each 28 day cycle
  Other Names: Tarceva
Drug: Maintenance erlotinib — 150 mg po daily (days 1 - 28 of 28 day cycle)
  Other Names: Tarceva

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving bendamustine together with erlotinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving bendamustine together with erlotinib in treating patients with stage IIIB, stage IIIC, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the phase II dose and assess the toxicity of bendamustine hydrochloride and erlotinib hydrochloride in patients with triple-receptor (estrogen receptor, progesterone receptor, and HER-2)-negative, stage IIIB, IIIC, or IV breast cancer. (Phase I)
* To determine the efficacy of this regimen in these patients. (Phase II)

Secondary (Correlative)

* To assess the correlation between tumor EGFR expression and EGFR gene amplification and treatment efficacy and toxicity.
* To assess for differences in treatment efficacy between basal-like and non-basal-like cancers.
* To assess for differences in treatment efficacy between tumors with and without expression of DNA damage-response (DDR) checkpoint proteins.
* To assess for differences in the activation state of DDR checkpoint proteins based on breast cancer subtype.

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II study.

Patients receive bendamustine hydrochloride IV over 30 minutes on days 1-2 and oral erlotinib hydrochloride once daily on days 5-21. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with no evidence of disease progression may continue with daily single-agent oral erlotinib hydrochloride on days 1-28. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Breast cancer tissue blocks from prior procedures are obtained for correlative studies. After a tissue microarray (TMA) and a TMA map are prepared, TMA slides are used for hematoxylin and eosin (H&E) staining, FISH, and IHC.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer meeting 1 of the following criteria:

  * Unresectable stage IIIB or IIIC disease
  * Stage IV disease
* Must be negative for all of the following:

  * Estrogen receptor (< 10%)
  * Progesterone receptor (<10%)
  * HER-2 (negative FISH, IHC 0 - 1+, or IHC +2 with negative FISH)
* Measurable or evaluable disease
* No symptomatic or progressive CNS (central nervous system) metastases

  * Previously treated CNS metastases allowed provided all of the following criteria are met:

    * At least 8 weeks since prior radiation to brain or CNS metastases
    * No concurrent steroids
    * No leptomeningeal disease

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Life expectancy ≥ 6 months
* WBC > 1,500/mm³
* Platelet count > 100,000/mm³
* Creatinine clearance > 40 mL/min
* Normal electrolytes (i.e., Na, K, and Ca normal; minor deviations are allowed if they do not impact on patient safety in the clinical judgment of the treating physician)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN in the presence of documented liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver or bone metastases)
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception
* No uncontrolled intercurrent illness
* No active infection requiring systemic therapy
* Able to swallow oral medications and with no medical problems or prior surgeries that may interfere with the absorption of oral medications including the following:

  * Uncontrolled nausea, vomiting, or diarrhea
  * Lack of the physical integrity of the upper gastrointestinal tract
  * Malabsorption syndrome
* No known hypersensitivity to bendamustine hydrochloride, mannitol, or erlotinib hydrochloride
* No prior malignancy in the past 5 years except for adequately treated basal cell or squamous cell skin carcinoma, or adequately treated stage I-II cancer for which the patient is in complete remission

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior adjuvant or neoadjuvant chemotherapy and 1 prior chemotherapy regimen in the metastatic setting allowed provided recovered from all acute toxicities
* No prior bendamustine hydrochloride or EGFR-directed therapy
* No other concurrent antineoplastic treatments, including radiotherapy, chemotherapy, biological therapy, hormonal therapy, immunotherapy, gene therapy, and surgery

  * Intravenous bisphosphonates allowed
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Layman, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Layman RM, Ruppert AS, Lynn M, Mrozek E, Ramaswamy B, Lustberg MB, Wesolowski R, Ottman S, Carothers S, Bingman A, Reinbolt R, Kraut EH, Shapiro CL. Severe and prolonged lymphopenia observed in patients treated with bendamustine and erlotinib for metastatic triple negative breast cancer. Cancer Chemother Pharmacol. 2013 May;71(5):1183-90. doi: 10.1007/s00280-013-2112-2. Epub 2013 Feb 21. PMID 23430121
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine and Erlotinib: Patients in dose level I were administered Bendamustine 100 or 120 mg/m2 IV on days 1 and 2 and 100 mg PO of Erlotinib on days 5 - 21 of each 28 day cycle.
Period: Overall Study
Arm/Group | Bendamustine and Erlotinib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 53 [38 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
ECOG (Eastern Cooperative Oncology Group) performance status [Number; unit: participants]
  0 (Fully active) | 4
  1 (Restricted) | 6
  2 (Ambulatory and capable selfcare) | 1
Site of metastasis [Number; unit: participants] — A patient can be represented among multiple sites
  participants
    Lymph nodes | 9
    Lung/pleura | 6
    Bone | 4
    Liver | 3
    Chest wall/skin | 3
    Brain | 1
Prior chemotherapy [Number; unit: participants]
  Adjuvant only | 4
  Metastasis/local recurrence only | 1
  Both | 6
Total number of prior treatment regimens [Number; unit: participants]
  1 prior regimen | 4
  2 prior regimens | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose of Bendamustine Hydrochloride (Phase I)
Description: 28 day cycle included intravenous bendamustine on days 1 and 2.
Time Frame: Up to two years
Measure: Number; unit: mg/m^2
Groups:
- Bendamustine and Erlotinib: Participants in dose level I were administered 100 mg/m^2 IV of Bendamustine on days 1 and 2 and 100 mg PO of Erlotinib on days 5 - 21 of each 28 day cycle.
  Participants in dose level II were administered 120 mg/m^2 IV of Bendamustine on days 1 and 2 and 150 mg PO of Erlotinib on days 5 - 21 of each 28 day cycle.
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
mg/m^2 | 120

2. Primary Outcome: Maximum-tolerated Dose of Erlotinib Hydrochloride (Phase I)
Description: 28 day cycle included intravenous erlotinib on days 15-21.
Time Frame: Up to two years
Measure: Number; unit: mg
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
mg | 150

3. Primary Outcome: Dose-limiting Toxicity (Phase I)
Time Frame: Up to two years
Measure: Number; unit: patients
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
patients
  Dose level I, n=5 | 0
  Dose level II, n=6 | 1

4. Primary Outcome: Progression-free Survival at 6 Months and 12 Months (Phase II)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to two years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
months | 3.7 [1.7 to 5.5]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to two years
Measure: Number; unit: patients
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
patients
  Dose Level 1 | 0
  Dose Level 2 | 1

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Time Frame: Up to two years
Population: The data was not collected and analyzed
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Response (DR)
Time Frame: Up to two years
Measure: Median (95% Confidence Interval); unit: months to progression
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
months to progression | 3.7 [1.7 to 5.5]

8. Secondary Outcome: Overall Survival (OS)
Time Frame: from time of study enrollment until death, for up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 11
months | 10.8 [3.6 to 13.1]

9. Secondary Outcome: Relationship of EGFR Expression or Amplification, Basal-like Tumors, and DNA Damage-repair Checkpoint Activation With ORR, CBR, DR, and OS
Time Frame: up to two years
Population: Correlative studies to assess EGFR expression and gene amplification, were planned, but not collected because of early trial termination.
Arm/Group | Bendamustine and Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from beginning of cycle 1 treatment through end of treatment, for up to 2 years
Description: This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0 for toxicity and Serious Adverse Event reporting.
Arm/Group | Bendamustine and Erlotinib
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine and Erlotinib (N=11)
Infection (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine and Erlotinib (N=11)
Leukopenia (Investigations) | 9 (9)
Neutropenia (General disorders) | 4 (4)
Lymphopenia (Investigations) | 11 (11)
CD4 count (Investigations) | 7 (7)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6)
Platelets (Investigations) | 7 (7)
Hypersensitivity (Immune system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 3 (3)
Consitutional (General disorders) | 7 (7)
Metabolic (Metabolism and nutrition disorders) | 6 (6)
Pulmonary (Cardiac disorders) | 4 (4)
Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No